CLINICAL TRIAL: NCT04118725
Title: Assessment of Muscular Respiratory Involvement in Systemic Sclerosis
Brief Title: Muscular Respiratory Involvement and Systemic Sclerosis
Acronym: SIROCO
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Poitiers University Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: 2019-A01047-50
Record Dates: First submitted 2019-09-26; First posted 2019-10-08 (Actual); Last update posted 2021-09-29 (Actual); Status verified 2021-09

CONDITIONS: Systemic Sclerosis; Diaphragm Defect; Respiratory Insufficiency; Pulmonary Function Test; Diaphragmatic Electromyography; Muscular Weakness
MeSH Terms: conditions — Scleroderma, Systemic; Respiratory Insufficiency; Muscle Weakness | interventions — Respiratory Function Tests

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Muscular explorations (Experimental): Pulmonary function test and diaphragmatic electromyography
  Interventions: Diagnostic Test: Pulmonary function test

INTERVENTIONS:
Diagnostic Test: Pulmonary function test — Diaphragmatic electromyography with measurement of transdiaphragmatic pressure in cases of dyspnea and/or abnormal pulmonary function test (maximum inspiratory pressure and/or lying/seating low vital capacity ratio)

SUMMARY:
Dyspnea in systemic sclerosis (ScS) constitute a major factor of functional disability.

Intensity of dyspnea is sometimes discordant with objectives data from cardiopulmonary involvements, suggesting unknown additional factors.

Diffuse fibrosing myopathy of bad prognosis have been reported in ScS.To now, muscular respiratory involvement has not been evaluated in ScS. Therefore, ScS patients (with or without dyspnea) could have underlying respiratory muscular involvement not detected by current standard of care with pulmonary function tests (PFT).

This project is the first, to the best of our knowledge, to assess frequency of respiratory muscular involvement in ScS and to evaluate a screening strategy of this involvement.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 years-old
* ScS fulfilling ACR/EULAR 2013 classification criteria and followed in the department of internal medicine of Poitiers University Hospital
* Written informatory consent

Exclusion Criteria:

* Individuals under tutorship or guardianship
* Individuals with reinforced protection: minors, judiciary or administrative decision
* No affiliation to social insurance
* Pregnancy or breastfeeding
* Associated neuromuscular disease (myasthenia, degenerative diseases)
* Bedridden individuals or with health condition not allowing realization or interpretation of PFT and/or EMG (acute cardiac and/or respiratory failure, pneumopathy)
* Individuals with pacemaker and implanted pumps, especially sensing dispositives, as defibrillators ( relative contre-indication to EMG with magnetic stimulation)
* Individuals with contre-indication to gastroesophageal probe: INR >4, oesophageal varices, suspected cardio-facial fracture, oesophageal and/or facial obstacle

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 52 (Actual)
Dates: Start 2019-10-21 (Actual); Primary Completion 2021-07-07 (Actual); Study Completion 2021-07-07 (Actual)

PRIMARY OUTCOMES:
Frequency of diaphragmatic involvement among ScS patients with dyspnea and/or with suspected respiratory muscular involvement on pulmonary function tests (PFT) | 4 months maximum (maximum time between PFT realization and date to obtain EMG/Pdi)
  Number of patients with dyspnea (SADOUL ≥2) and/or with respiratory muscular involvement suspected on PFT (maximum inspiratory pressure (max IP) below definite z-score and/or lying/sitting low vital capacity (LVC) ratio < 75%) having diaphragmatic muscular involvement confirmed by diaphragmatic electromyography (EMG) (latency >8.5ms and amplitudes <0.5mV) by neck electric phrenic stimulation and/or Pdi <20cmH2O after magnetic stimulation

SECONDARY OUTCOMES:
Sensitivity, specificity, positive and negative predictive value of pulmonary function tests compared to diaphragmatic involvement confirmed by EMG and Pdi among ScS patients with suspected pulmonary muscular involvement on PFT | 4 months maximum (maximum time between PFT realization and date to obtain EMG/Pdi)
  Proportion of ScS patients with diaphragmatic involvement confirmed by EMG (latency >8.5ms and amplitudes <0.5mV by neck electric phrenic stimulation and/or Pdi <20cmH2O after magnetic stimulation) compared to proportion of ScS patients with maxIP below definite z-score and/or lying/sitting LVC ratio <75%
Sensitivity, specificity, positive and negative predictive value of dyspnea compared to diaphragmatic involvement confirmed by EMG and Pdi | 4 months maximum (maximum time between PFT realization and date to obtain EMG/Pdi)
  Proportion of ScS patients with diaphragmatic involvement confirmed by EMG (latency >8.5ms and amplitudes <0.5mV by neck electric phrenic stimulation and/or Pdi <20cmH2O after magnetic stimulation) compared to proportion of ScS patients with dyspnea (SADOUL ≥2) or without dyspnea
Correlation between diaphragmatic involvement confirmed by EMG and and/or Pdi and dyspnea | 4 months maximum (maximum time between PFT realization and date to obtain EMG/Pdi)
  Proportion of ScS patients with diaphragmatic involvement confirmed by EMG (latency >8.5ms and amplitudes <0.5mV by neck electric phrenic stimulation and/or Pdi <20cmH2O after magnetic stimulation) and proportion of ScS patients with dyspnea (SADOUL ≥2)
Correlation between diaphragmatic involvement confirmed by EMG and and/or Pdi and general and ScS-related factors | 4 months maximum (maximum time between PFT realization and date to obtain EMG/Pdi)
  Proportion of ScS patients with diaphragmatic involvement confirmed by EMG (latency >8.5ms and amplitudes <0.5mV by neck electric phrenic stimulation and/or Pdi <20cmH2O after magnetic stimulation) and : age in years ; proportion of female; proportion of limited cutaneous or diffuse cutaneous or sine scleroderma ; ScS duration in years, proportion of anti-centromere or anti-Scl70 or anti-ARNpolymeraseIII or "others" autoantibody; proportion of digital tip ulcerations; proportion of subcutaneous calcifications; proportion of arthritis; proportion of arterial pulmonary hypertension; proportion of interstitial lung disease; proportion of renal crisis; proportion of inflammatory myopathy; proportion of immunosuppressant use; modified Rodnan skin score (median, ranging from 0-51)); interlabial length in centimeter; proportion of telangiectasia; proportion of cardiac insufficiency (left and/or right heart); creatine phosphokinase level in UI/mL ; PO2 in mmHg; PCO2 in mmHg
Correlation between diaphragmatic involvement confirmed by EMG and and/or Pdi and suspected muscular respiratory on pulmonary function test | 4 months maximum (maximum time between PFT realization and date to obtain EMG/Pdi)
  Proportion of ScS patients with diaphragmatic involvement confirmed by EMG (latency >8.5ms and amplitudes <0.5mV by neck electric phrenic stimulation and/or Pdi <20cmH2O after magnetic stimulation) and proportion of patients with maxIP below definite z-score and/or lying/sitting LVC ratio < 75%)
Correlation between diaphragmatic involvement confirmed by EMG and and/or Pdi and quality of life and functional disability | 4 months maximum (maximum time between PFT realization and date to obtain EMG/Pdi)
  Proportion of ScS patients with diaphragmatic involvement confirmed by EMG (latency >8.5ms and amplitudes <0.5mV by neck electric phrenic stimulation and/or Pdi <20cmH2O after magnetic stimulation) and total score in the Functional Assessment of Chronic Illness Therapy (FACIT)-Dyspnea-short form (ranging from 0 to 30; higher values represent a worse outcome); physical summary score (mean) from the short form health survey 36 (SF-36) (French version 2.0) ranging from 0 to 100 (higher values represent a worse outcome) ; mental summary score (mean) from the short form health survey 36 (SF-36) (French version 2.0) ranging from 0 to 100 (higher values represent a worse outcome

CONTACTS AND LOCATIONS:
Locations (1):
- Chu de Poitiers, Poitiers, France

IPD SHARING:
Plan to Share IPD: Undecided